CLINICAL TRIAL: NCT00791232
Title: A Randomized, Double-blind, Placebo- and Active-controlled, Parallel-group, Phase 1 Study to Compare the Tolerability of OROS Paliperidone (Extended Release) With Immediate-release (IR) Risperidone in Subjects With Schizophrenia
Brief Title: A Study of Extended Release Extended-release (ER) OROS Paliperidone Tolerability, as Compared to Immediate-release (IR)Risperidone, in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004273
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Extended-release paliperidone; Schizophrenia, Mood disorders, Antipsychotic drugs; ER OROS paliperidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders

INTERVENTIONS:
Drug: extended-release (ER) OROS paliperidone

SUMMARY:
The purpose of this study is a noninferiority comparison of the orthostatic tolerability of a dose of 12 mg extended-release (ER) OROS paliperidone with the current recommended initial titration dose (2 mg) of immediate-release (IR) risperidone in patients with schizophrenia. Other study objectives are 1) to compare the tolerability and safety of a clinically equivalent fixed dose of ER OROS paliperidone with the currently recommended dose of risperidone, 2) to compare the early tolerability of the 2 treatments with placebo, 3) to compare tolerability of the 2 treatments, using a population pharmacokinetic/pharmacodynamic (pop PK/PD) model, to 4) assess the relationship between genetic variability in drug metabolizing enzymes and interindividual variability in plasma exposure to paliperidone or risperidone within each treatment group.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo- and active-controlled, parallel group, Phase 1. The study in patients with schizophrenia consists of a 1 week, open-label, placebo washout period (Days -7 to -1) and a 6 day double-blind treatment period during which patients will receive 1 of 3 treatments: placebo on Day 1 and ER OROS paliperidone (12 mg) on Days 2 to 6, ER OROS paliperidone (12 mg) on Days 1 to 6, or IR risperidone 2 mg on Day 1 and 4 mg on Days 2 to 6. Safety and tolerability will be monitored throughout the study.. ER OROS paliperidone (12 mg, oral) on Days 2 to 6, ER OROS paliperidone (12 mg, oral) on Days 1 to 6, or IR risperidone (oral) 2 mg on Day 1 and 4 mg on Days 2 to 6

ELIGIBILITY:
Inclusion Criteria:

* Willingness to spend 2 weeks as an in-patient during the washout and treatment period
* Currently treated with oral risperidone antipsychotic monotherapy for at least 1 month prior to screening
* DSM-IV diagnosis of schizophrenia (Patients with a diagnosis of schizophrenia [paranoid type (295.30), disorganized type (295.10), catatonic type (295.20), undifferentiated type (295.90), or residual type (295.60)] as defined by DSM-IV criteria
* Absence of acute exacerbation for a minimum of 6 months prior to screening
* Female patients must be postmenopausal for at least 1 year, surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before screening and throughout the study, and have a negative urine pregnancy test at screening and baseline
* The patient is otherwise healthy on the basis of a physical examination, medical history, electrocardiogram, and the results of blood biochemistry and hematology tests and a urinalysis performed within 30 days of the start of the treatment period. If the results of the biochemistry or hematology tests or the urinalysis testing are not within the laboratory's reference ranges, the patient may be included only on condition that the investigator judges that the deviations are not clinically significant.

Exclusion Criteria:

* Involuntarily committed in-patients
* Patients who have received long-acting depot antipsychotic medication (discontinued RISPERDAL CONSTA for less than 10 weeks or discontinued other depots for less than 2 cycles)
* Any significant history of cardiovascular disease: atrial fibrillation or flutter, second and third degree heart block and equivalent, resting supraventricular tachycardia (>100 beats per minute), unstable atherosclerotic heart disease, valvular abnormality
* Body Mass Index > = 35 kg/m2 or a history of or current hypertension
* Use of disallowed concomitant therapy or patients likely to require prohibited concomitant therapy during participation in the study
* Patients with a pacemaker
* Concomitant disease of the central nervous system that would bias the study evaluations, e.g.
* stroke, brain tumor, Parkinson's disease, significant brain trauma, Alzheimer's disease, epilepsy, multiple sclerosis, currently-treated migraine
* A DSM-IV Axis I diagnosis other than schizophrenia or with a DSM-IV diagnosis of substance dependence within 6 months prior to screening evaluation (nicotine and caffeine dependence are not exclusionary)
* Diabetes mellitus and/or repeated fasting blood glucose value during the washout period >126 mg/dl and /or HbA1C > 7. 5%, hypothalamo-hypophyse dysfunction, Cushing, Addison, thyrotoxicosis, or Anemia (as defined by hematocrit < 30%)
* Suicidal or homicidal ideation
* Positive drug screen at screening and at baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2003-03; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
A non-inferiority comparison of the orthostatic tolerability of a higher initial dose of paliperidone OROS with the current recommended initial dose of risperidone in patients with schizophrenia

SECONDARY OUTCOMES:
To compare the tolerability and safety of a clinically equivalent fixed dose of paliperidone OROS with the recommended dose of risperidone; early tolerability of the two formulations with placebo; tolerability using a pop PK/PD model

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of ER OROS paliperidone tolerability, as compared to IR risperidone, in patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=576&filename=CR004273_CSR.pdf